CLINICAL TRIAL: NCT05470738
Title: PAncreas Borderline and Locally Advanced Snapshot Study
Acronym: PALASS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2022 GAGNIERE PALASS
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; adenocarcinoma; locally advanced cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project's objective is to carry out prospectively, in France, for one year, a descriptive registry study in the management of patients with borderline or locally advanced pancreatic adenocarcinoma, and to collect both the patient's demographic characteristics, but also the therapeutic regimens applied, the types of surgeries performed and the outcome of the patients after surgery, and at three months of follow up (preoperative data, complications's post surgery, quality of the resection, etc.)

DETAILED DESCRIPTION:
* Multicenter, observational prospective study over one year in France in patients with borderline or locally advanced pancreatic adenocarcinoma operated between September 2022 and August 2023.
* Patients will be screened by the pancreatic's surgeons practicing in a reference centers during preoperative surgical consultations (V1),
* The patient's non-objection will be sollected,
* The end of follow-up's patient will take place during the post-operative consultation approximately 3 months after surgery (V3)
* Between V1 and V3, preoperative data (demography, history, tumor characteristics, neoadjuvant treatments performed, tumor response), operative, intraoperative, pathological and postoperative data will be collected via a e-CRF " the REDCAP software".

ELIGIBILITY:
Inclusion Criteria:

* Any patient over the age of 18, operated on for pancreatic adenocarcinoma, borderline or locally advanced, between September 2022 and August 2023, in France
* Diagnosis of pancreatic adenocarcinoma:

  * either after cytopuncture with anatomopathological result confirming the diagnosis,
  * or with strong suspicion on the combined criterias : clinical, biological and morphological criterion (according to INCa 2019 and NCCN recommendations ) in the event of absence of anatomopathological documentation (failure of several fine needle punctures (maximum 3)/or non-contributory anatomopathological examinations),
* Borderline or locally advanced character depending on the presence of a contact of the tumor with nearby vessels and defined by morphological examination (scanner +/- MRI). These criteria are defined by the NCCN Guidelines for Pancreatic Adenocarcinoma V.1.2021, international reference

Exclusion Criteria:

* Patient under juridic protected or subject to any measure of legal protection,
* Patients not operated on for their pancreatic adenocarcinoma,
* Adenocarcinoma of the pancreas operable immediately on diagnosis,
* Metastatic pancreatic adenocarcinoma from the outset on diagnosis,
* Patient without pancreatic adenocarcinoma after histological examination (in the case where the pancreatic lesion was operated on for strong suspicion of pancreatic adenocarcinoma on the combined clinical, biological and morphological criterion (according to INCa 2019 and NCCN recommendations, but that the lesion on definitive pathological examination is not a pancreatic adenocarcinoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient operated on for pancreatic adenocarcinoma, borderline or locally advanced, between September 2022 and August 2023, in France
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2023-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
The main study's objective is to definite the effective rate of adjuvant chemotherapy performed after surgery (at the 3-month post operatively), which is essential marker recognized as improving overall survival. | during 1 year
  Evaluation of the rate of adjuvant chemotherapy performed after surgery (at the 3-month post operatively)

SECONDARY OUTCOMES:
The secondary objective of the study is to know, in patients operated for pancreatic adenocarcinoma, the rate of postoperative complications, the rate of the postoperative morbidity and mortality, and the quality of the resection. | during 1 year
  the secondary objective will be definited by evaluation of the rate of postoperative complications, the rate of postoperative morbidity and mortality and the quality of the resection (R0)

CONTACTS AND LOCATIONS:
Overall Officials: Johan Gagniere, Study Director — University Hospital, Clermont-Ferrand
Locations (23):
- France (23):
  - CHU Amiens, Amiens
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHU clermont-ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHU Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - APHM, Marseille
  - Institut Paoli-Calmettes d'Unicancer, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - APHP Hopital Beaujon, Paris
  - APHP Hopital Cochin, Paris
  - APHP Hopital de la Pitié-Salpétrière, Paris
  - APHP Hopital Paul Brousse, Paris
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No